CLINICAL TRIAL: NCT06744764
Title: Pulsed Electromagnetic Fields in Preventing Physical Deconditioning in Patients Undergoing Prolonged Hospitalization: A Case Match Control Study
Brief Title: Pulsed Electromagnetic Fields in Preventing Physical Deconditioning in Patients Undergoing Prolonged Hospitalization
Acronym: PEMF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2022/00928
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Haematological Cancer; Healthy
Keywords: Magnetic therapy; Cancer management; Muscle atrophy
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Clinical trial coordinators
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Haematology Patients (Experimental): Patients will receive 1mT magnetic therapy twice per week for 4 consecutive weeks.
  Interventions: Device: PEMF (1mT)
- Haematology Patients (Case-matched) (No Intervention): Case-matched haematology patients will be recruited after 20 haematology patients receiving the intervention has been recruited. The parameters for matching would be chemotherapy vs bone marrow transplant, age and fitness level according to the short physical performance battery (SPPB) score (0-2, 3-9, 10-12).
- Healthy Volunteers (PEMF) (Experimental): Healthy volunteers will receive 1mT magnetic therapy twice per week for 4 consecutive weeks.
  Interventions: Device: PEMF (1mT)
- Healthy volunteers (Sham) (Sham Comparator): Healthy volunteers will place their legs in the PEMF device, same as the volunteers receiving the therapy, twice per week for 4 consecutive weeks. However, no magnetic stimulation will be given to this group.
  Interventions: Device: PEMF (0mT)

INTERVENTIONS:
Device: PEMF (1mT) — 1mT of field strength will be given to patients/healthy volunteers for 10 minutes, twice per week for 4 consecutive weeks.
  Arms: Haematology Patients; Healthy Volunteers (PEMF)
Device: PEMF (0mT) — Healthy volunteers will place their legs in the PEMF device, twice per week for 4 consecutive weeks. However, no magnetic stimulation will be given.
  Arms: Healthy volunteers (Sham)

SUMMARY:
The goal of this clinical trial is to examine if pulsed electromagnetic fields (PEMF) can prevent or decrease physical deconditioning associated with prolonged hospitalisation and immobility of haematology patients. The main question[s] it aims to answer [is/are]:

* Does haematology patients undergoing prolonged hospitalisation have no or decreased physical deconditioning when exposed to PEMF?
* What are the changes in muscle secretome at baseline and after exposure to PEMF? Researchers will compare haematology patients who receive PEMF against patients who did not receive the treatment to see if there is a change in physical deconditioning. Healthy volunteers will also be recruited and randomized to either exposure to PEMF or no exposure.

Haematology patients will

* Have their blood taken at baseline, 4 weeks from baseline and 8 weeks from baseline.
* Undergo SPPB test at baseline, 4 weeks and 8 weeks from baseline, and the test comprises of the time up and go test, 4 minute walk test and sit to stand test.
* Either expose to PEMF twice per week for 4 consecutive weeks or no exposure. Healthy volunteers will
* Have their blood taken at baseline, 4 weeks from baseline and 8 weeks from baseline.
* Either expose to PEMF twice per week for 4 consecutive weeks or no exposure.

ELIGIBILITY:
Inclusion Criteria:

* Haematology patients who are undergoing induction chemotherapy for acute leukemia
* Haematology patients who are undergoing haematopoietic stem cell transplant
* Have ECOG 0-24. Able to walk at baseline to participate in short physical battery test.
* For healthy volunteers, subjects have to be healthy without any major disease states, not on any drugs or requiring long term medical attention.

Exclusion Criteria:

* Patients who do not agree to sign the consent form.
* Pregnant women will be excluded from the study for healthy volunteers

Ages: 25 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in physical deconditioning in haematology patients after 8 sessions of PEMF | Change in SPPB test result 4 and 8 weeks from baseline
  The haematology patients will undergo the SPPB test which comprises of the time up and go (TUG) test, 4 minute walk test and 5 times sit to stand (STS) test. The same test will be repeated 4 and 8 weeks from baseline. Based on the case study report done previously, we anticipate an improvement of TUG mean by 1.9sec, 5-times STS by 2.3sec and 4 min walk test by 0.14meters by the end of the 8 week therapy. We will consider the trend to be significant if 2 out of 3 three parameters in the SPPB are met.
Changes in the levels of anti-cancer factors in blood plasma from haematology patients and healthy volunteers | Change in anti-cancer biomarkers levels in blood plasma from PEMF-exposed patients at week 4 and week 8 versus their own baseline.
  Anti-cancer factors such as HTRA1 and Klotho can be altered with PEMF therapy in humans.

CONTACTS AND LOCATIONS:
Locations (2):
- Singapore (2):
  - NUHS Investigational Medicine Unit, Kent Ridge
  - National University Hospital, Kent Ridge

IPD SHARING:
Plan to Share IPD: Yes
Age, ethnicity, medical history, diet, physical activity, anthropometrics
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Venugobal S, Tai YK, Goh J, Teh S, Wong C, Goh I, Maier AB, Kennedy BK, Franco-Obregon A. Brief, weekly magnetic muscle therapy improves mobility and lean body mass in older adults: a Southeast Asia community case study. Aging (Albany NY). 2023 Mar 19;15(6):1768-1790. doi: 10.18632/aging.204597. Epub 2023 Mar 19. PMID 36934330
- [Background] Stephenson MC, Krishna L, Pannir Selvan RM, Tai YK, Kit Wong CJ, Yin JN, Toh SJ, Torta F, Triebl A, Frohlich J, Beyer C, Li JZ, Tan SS, Wong CK, Chinnasamy D, Pakkiri LS, Lee Drum C, Wenk MR, Totman JJ, Franco-Obregon A. Magnetic field therapy enhances muscle mitochondrial bioenergetics and attenuates systemic ceramide levels following ACL reconstruction: Southeast Asian randomized-controlled pilot trial. J Orthop Translat. 2022 Oct 13;35:99-112. doi: 10.1016/j.jot.2022.09.011. eCollection 2022 Jul. PMID 36262374
- [Background] Yap JLY, Tai YK, Frohlich J, Fong CHH, Yin JN, Foo ZL, Ramanan S, Beyer C, Toh SJ, Casarosa M, Bharathy N, Kala MP, Egli M, Taneja R, Lee CN, Franco-Obregon A. Ambient and supplemental magnetic fields promote myogenesis via a TRPC1-mitochondrial axis: evidence of a magnetic mitohormetic mechanism. FASEB J. 2019 Nov;33(11):12853-12872. doi: 10.1096/fj.201900057R. Epub 2019 Sep 13. PMID 31518158
- [Derived] Iversen JN, Tai YK, Yap JLY, Abdul Razar RBB, Sukumar VK, Wu KY, Ooi MG, Kukumberg M, Adam S, Rufaihah AJ, Franco-Obregon A. One Month of Brief Weekly Magnetic Field Therapy Enhances the Anticancer Potential of Female Human Sera: Randomized Double-Blind Pilot Study. Cells. 2025 Feb 23;14(5):331. doi: 10.3390/cells14050331. PMID 40072060

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2024-04-11): https://cdn.clinicaltrials.gov/large-docs/64/NCT06744764/Prot_ICF_000.pdf